CLINICAL TRIAL: NCT05237076
Title: Carotid Body Dysfunction in Type 2 Diabetes
Brief Title: Carotid Body Function in Type 2 Diabetes Mellitus
Acronym: CBHypoxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Demcon (Industry)
Responsible Party: Principal Investigator, Albert Dahan, Principal Investigator, Leiden University Medical Center
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: NL78476.058.21
Record Dates: First submitted 2022-02-02; First posted 2022-02-11 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Diabetes Mellitus, Type 2; Hypoxia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypoxia

STUDY DESIGN:
Intervention Model Description: Multi arm pre-post study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetes Type 2 (Experimental): Patients with DM Type 2 using Oral Diabetes Medications only.
  Interventions: Diagnostic Test: Hyperinsulemic-Euglycemic Clamp & Hypoxic Ventilatory Response (HVR)
- Healthy controls (Active Comparator): Healthy controls without comorbidities.
  Interventions: Diagnostic Test: Hyperinsulemic-Euglycemic Clamp & Hypoxic Ventilatory Response (HVR)

INTERVENTIONS:
Diagnostic Test: Hyperinsulemic-Euglycemic Clamp & Hypoxic Ventilatory Response (HVR) — Hyperinsulemic-Euglycemic Clamp as described by deFronzo et al.

SUMMARY:
This trial will assess chemosensitivity differences of the carotid bodies in individuals with T2DM, compared to healthy controls. During baseline and hyperinsulinemia.

DETAILED DESCRIPTION:
During the COVID-19 pandemic patients with comorbidities such as hypertension, diabetes mellitus, obesity and pregnancy were overrepresented in the population that was admitted to the hospital. Morbidity and mortality due to SARS-COV-2 infection was higher in these patients compared to patients without these comorbidities. The higher incidence, morbidity and mortality is suggestive of an underlying mechanism that puts these patients more at risk. A proposed mechanism is the sympathetic overactivity that is associated with these conditions. Recently, it has become clear that the carotid bodies play an important role in sympathetic overactivity in these conditions. Dysfunction of this organ is associated with decreased chemosensitivity, disruption of insulin sensitivity, but is also associated with changes in neurohumoral control in response to infection. Whether carotid body dysfunction can explain the severity of SARS-COV-2 infection remains to be seen. The aim of this study is to find whether patients with type 2 diabetes have altered chemosensitivity and are in fact sympathetically overactive compared to healthy controls and during a hyperinsulinemic-euglycemic clamp. Findings could help explain why type 2 diabetes patients are more heavily affected by SARS-COV-2 and could identify potential targets for treatment in these patients.

ELIGIBILITY:
Inclusion criteria

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* 18 years and older
* Subjects must be willing to give written informed consent for the trial and able to adhere to dose and visit schedule.
* Non-insulin-dependent diabetes mellitus (NIDDM) or healthy sex, age (± 3 yrs) and BMI (± 3 kg/m2) matched controls.
* Have no clinical or electrocardiographic signs of ischemic heart disease as determined by the Investigator with normal cardiac intervals appropriate for their gender. The Screening 12 lead ECG conduction intervals must be within gender specific normal range (e.g., QTcF ≤ 430 msec, PR interval ≤ 220 msec). ECGs are to be judged by the investigator or sub investigator as per standardized procedures.
* Vital sign measurements must be within the following ranges: (Individuals with values outside (or indicate lower or higher) of these ranges may be enrolled if clinically acceptable to the investigator and sponsor.

  * body temperature, between 35.5°C and 37.5°C
  * systolic blood pressure, 90 to 150 mmHg
  * diastolic blood pressure, 40 to 95 mmHg
  * pulse rate, 40 to 100 bpm
* Subjects must be free of any clinically significant disease that would interfere with the study evaluations.
* Subjects presenting out of range values of lab/ECG/vital signs compatible with normal variation of the normal healthy subject can be included in the study at the investigator's discretion and sponsor written approval.
* Positive Allen's test
* Fitzpatrick skin type I or II

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Insulin dependent diabetes mellitus
* Diagnosed Obstructive Sleep Apnea (OSAS) or high suspicion of OSAS determined by a STOP-BANG score > 5
* Respiratory or cardiovascular disease
* Smoking/vaping
* Positive pregnancy test
* conditions that result in elevated levels of methaemoglobinia
* body mass index > 35 kg/m2
* Use of illicit drugs
* Use of prescription opioids or benzodiazepines
* Failure of the drug of abuse tests at screening or check-in.
* History of dyspnea, asthma, tuberculosis, chronic obstructive pulmonary disease, or any other ventilatory / lung disease.
* Subjects with excessive facial hair preventing sealing of the occlusive face mask.
* Subjects who, in the opinion of the investigator, will not be able to participate optimally in the study.
* Subject who has a history of any infectious disease within 4 weeks prior to drug administration that in the opinion of the investigator, affects the subject's ability to participate in the trial.
* Subjects who are part of the study staff personnel or family members of the study staff personnel.
* Subjects who have demonstrated allergic reactions (e.g., food, drug, atopic reactions or asthmatic episodes) which, in the opinion of the investigator and sponsor, interfere with their ability to participate in the trial.
* Personal or family history of arrhythmias or ECG conductance abnormalities.
* Hypokalemia defined as <3.5 mmol/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Chemosensitivity of carotid bodies during baseline and euglycemic clamp | 5 minutes
  L/min/PaO2

SECONDARY OUTCOMES:
HRV during baseline and euglycemic clamp | 30 min
  HRV parameters

CONTACTS AND LOCATIONS:
Overall Officials: Albert Dahan, MD, PhD, Principal Investigator — LUMC
Locations (1):
- LUMC, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
On request.